CLINICAL TRIAL: NCT01509144
Title: Phase 1, Randomised, Single-centre, Observer-blind Clinical Trial of Safety and Immunogenicity of Nasal-prime and Intramuscular Boost Immunisation With EN41-FPA2 HIV Vaccine in Healthy Female Volunteers
Brief Title: EuroNeut41: Safety & Immunogenicity of Immunisations With HIV Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PX'Therapeutics (Industry)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2010-023693-39
Record Dates: First submitted 2012-01-04; First posted 2012-01-12 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: HIV
Keywords: Safety of this HIV vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- nasal active low dose + IM active (Active Comparator): Group 1 Nasal vaccine - Low-dose (20 µg in 40 µL) IM vaccine (200 µg in 400 µL)
  Interventions: Biological: EN41-FPA2 HIV vaccine
- nasal active mid dose + IM active (Active Comparator): Group 2 Nasal vaccine - Mid-dose (100 µg in 200 µL) IM vaccine (200 µg in 400 µL)
  Interventions: Biological: EN41-FPA2 HIV vaccine
- nasal active full dose + IM active (Active Comparator): Group 3 Nasal vaccine - Full-dose (200 µg in 400 µL) IM vaccine (200 µg in 400 µL)
  Interventions: Biological: EN41-FPA2 HIV vaccine
- nasal placebo + IM active (Active Comparator): Group 4 Nasal Placebo - 400 µL IM vaccine (200 µg in 400 µL)
  Interventions: Biological: EN41-FPA2 HIV vaccine
- nasal placebo + IM placebo (Placebo Comparator): Group 5 Nasal placebo - 40 µL in Cohort 1 / 200 µL in Cohort 2 IM placebo (400 µL)
  Interventions: Biological: Na Cl Placebo vaccine

INTERVENTIONS:
Biological: EN41-FPA2 HIV vaccine — Group 1 Nasal vaccine - Low-dose (20 µg in 40 µL) IM vaccine (200 µg in 400 µL)
  Arms: nasal active low dose + IM active
Biological: EN41-FPA2 HIV vaccine — Group 2 Nasal vaccine - Mid-dose (100 µg in 200 µL) IM vaccine (200 µg in 400 µL)
  Arms: nasal active mid dose + IM active
Biological: EN41-FPA2 HIV vaccine — Group 3 Nasal vaccine - Full-dose (200 µg in 400 µL) IM vaccine (200 µg in 400 µL)
  Arms: nasal active full dose + IM active
Biological: EN41-FPA2 HIV vaccine — Group 4 Nasal Placebo - 400 µL IM vaccine (200 µg in 400 µL)
  Arms: nasal placebo + IM active
Biological: Na Cl Placebo vaccine — Group 5 Nasal placebo - 40 µL in Cohort 1 / 200 µL in Cohort 2 IM placebo (400 µL)
  Arms: nasal placebo + IM placebo

SUMMARY:
Objectives:

* To assess the safety of three priming immunisations by nasal route followed by two booster immunisations by intramuscular route
* To assess immunogenicity responses induced by the vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged between 18 and 55 years on the day of screening
2. Available for a maximal study duration of 12/13 months from the inclusion
3. Willing and able to give written informed consent
4. At low risk of HIV infection and willing to remain so for the duration of the study defined as:

   * no history of injecting drug use in the previous ten years
   * no gonorrhoea or syphilis in the last six months
   * no high risk partner (e.g. injecting drug use, HIV positive partner) either currently or within the past six months
   * no unprotected anal intercourse in the last six months, outside a relationship with a regular partner known to be HIV negative
   * no unprotected vaginal intercourse in the last six months outside a relationship with a regular known HIV negative partner
   * not had unprotected sex with someone from a region where HIV is more common (e.g Sub-Saharan African, Caribbean, South East Asia) outside a relationship with a regular known HIV negative partner
5. Negative HIV 1/2 antibody/antigen test at screening
6. If heterosexually active female, using an effective method of contraception with partner (combined oral contraceptive pill; injectable or implanted contraceptive; use of condoms incorporating spermicide if using these; physiological or anatomical sterility) from 14 days prior to the first vaccination until 6 months after the last, and willing to undergo urine pregnancy tests prior to each vaccination and blood pregnancy test at screening and final follow up.
7. Agree, to abstain from medications or other agents that are applied via the nasal route from 24 hours prior to each nasal vaccine dosing through to the safety assessment 1week later
8. Agree to abstain from donating blood during their participation in the trial
9. Registered with GP and medical history available for 12 months before dosing
10. Satisfactory response received from General Practitioner relating to medical history before randomization.

Exclusion Criteria:

1. Pregnant or lactating, or planning to get pregnant within the next year
2. Positive alcohol test
3. Positive drugs of abuse test
4. Clinically relevant abnormality on history or examination:

   * central nervous system disorder or disease, including
   * history of grand-mal epilepsy
   * cranial nerve palsies
   * severe eczema
   * severe epistaxis requiring surgical intervention or blood transfusion
   * clinically significant liver disease
   * clinically significant haematological, metabolic, gastrointestinal, renal, psychiatric or cardio-pulmonary disorders
   * ongoing infection;
   * autoimmune disease, immunodeficiency or use of immunosuppressive agents in preceding 3 months prior to dosing
   * using inhaled cortico-steroids and intranasal medications
5. Known or suspected history of clinically relevant nasal surgery, injury, nasal polyps or cleft palate, or a condition likely to require regular intranasal medication, which in the opinion of the investigator might interfere with intranasal vaccine administration
6. Known hypersensitivity to any component of the vaccine formulations used in this trial or have severe or multiple allergies
7. History of severe local or general reaction to vaccination defined as

   * local: extensive, indurated redness and swelling involving most of the antero-lateral thigh or the major circumference of the arm, not resolving within 72 hours
   * general: fever > 39.5°C within 48 hours; anaphylaxis; bronchospasm; laryngeal oedema; collapse; convulsions or encephalopathy within 72 hours
8. Receipt of live attenuated vaccine within 60 days or other vaccine within 14 days of scheduled study vaccine dosing
9. Receipt of an experimental vaccine containing HIV envelope proteins at any time in the past
10. Receipt of blood products or immunoglobin within 4 months of screening
11. Participation in another trial of a medicinal product, completed less than 90 days prior to Visit 2 and planned participation in another clinical trial during the present trial
12. HIV 1/2 antibody/antigen positive or indeterminate on screening
13. Positive for hepatitis B surface antigen, hepatitis C antibody or serology indicating active syphilis requiring treatment
14. Clinically significant routine laboratory parameters.
15. Unable to read and speak English to a fluency level adequate for the full comprehension of procedures required in participation and consent.
16. Unlikely to comply with protocol
17. History of drug or alcohol abuse or regular using of drugs, or who test positive in drugs of abuse and alcohol test at screening or admission
18. Has a condition, or is on regular medication (other than paracetamol, multivitamin, E45, or over the counter remedies) which in the opinion of the investigator is not suitable for participation in the study
19. Any local vaginal, cervical or gynaecological condition which may interfere with collection or interpretation of data collected through vaginal samples.
20. Using any Intra Uterine Contraceptive Device; as there is a risk of dislodging, displacing or removing the device when pulling or removing Softcup used for vaginal sampling.
21. Clinically significant abnormality on ECG performed at the screening visit
22. Any condition that, in the investigator's opinion, compromises the volunteer's ability to meet protocol requirements or to complete the study.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
• Safety of 5 EN41-FPA2 immunisations Primary Endpoints: AEs and IgG and IgA responses to EN41-FPA2 | up to 28 days after the final immunisation
  •Safety - Grade 3 or above adverse event. Any grade of adverse event that results in a clinical decision to discontinue further immunisations - Any grade of adverse event that occurs in a volunteer that has received at least one immunisation • Immunogenicity: Proportion of individuals mounting a serum IgG response to EN41-FPA2 at any time point up to 28 days after the final immunisation with 3 fold increase from pre-immunisation baseline sample taken at visit 2, week 0, priming #1. If no serum sample is available at this time point, serum taken at visit 1, screening may be substituted."

CONTACTS AND LOCATIONS:
Locations (1):
- Surrey Clinical Research Centre University of Surrey, Guildford, Surrey, United Kingdom